CLINICAL TRIAL: NCT07187752
Title: A Prospective and Multicenter Clinical Study to Identify the Molecular Characterization and Subtypes in Patients With HER2-positive Breast Cancer Receiving Neoadjuvant Trastuzumab and Pertuzumab.
Brief Title: Identification of HER2-Positive Breast Cancer Molecular Characterization and Subtypes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, PhD, MD, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-BC-QUPA-RWS-001
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Long-Term Synaptic Depression; pertuzumab; Drug Therapy; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab+Pertuzumab+Chemotherapy (Experimental): Participants will be administered at least 4-6 cycles of neoadjuvant pertuzumab plus trastuzumab -containing regimens chosen by the investigators prior to surgery.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Chemotherapy; Procedure: Excision of tumor/mastectomy

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab (8 mg/kg loading dose, followed by 6 mg/kg every 3 weeks)
  Other Names: QL1701 (A trastuzumab biosimilar produced by Qilu Pharmaceutical Co., Ltd)
Drug: Pertuzumab — Pertuzumab (loading dose 840 mg, followed by 420 mg every 3 weeks)
  Other Names: QL1209 (A pertuzumab biosimilar produced by Qilu Pharmaceutical Co., Ltd)
Drug: Chemotherapy — Chemotherapy chosen by the investigators.
Procedure: Excision of tumor/mastectomy — Definitive breast cancer surgery (excision or mastectomy) marks the end of protocol mandated therapy.

SUMMARY:
This study will evaluate the safety and efficacy of neoadjuvant trastuzumab, pertuzumab and chemotherapy chosen by the investigators and identify the molecular characterization and subtypes in human epidermal growth factor receptor 2 (HER2)-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years;
2. Eastern Cooperative Oncology Group (ECOG) score status 0-1.
3. Histologically confirmed invasive breast carcinoma with a primary tumor size of more than (>) 2 centimeters (cm) by standard local assessment technique; Breast cancer stage at presentation: early-stage (T2-3, N0-1, M0) or locally advanced (T2-3, N2 or N3, M0; T4, any N, M0);
4. HER2-positive breast cancer confirmed by immunohistochemistry or HER2 gene amplification by in situ hybridization;
5. Known estrogen receptor (ER) and progesterone receptor (PgR) status.
6. Has adequate bone marrow, renal, hepatic and blood clotting functions.
7. Left ventricular ejection fraction (LVEF) ≥50 percent (%).
8. Women of childbearing potential and men with partners of childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and after the last dose for at least 7 months. Negative serum or urine pregnancy test within 7 days before study enrollment.
9. Willing to provide tissue for research purposes.
10. Volunteer to participate in this study and sign the informed consent.

Exclusion Criteria:

1. Patients with stage IV metastatic breast cancer.
2. Bilateral invasive breast cancer;
3. Patients with breast cancer who have previously received anti-tumor therapy.
4. Occurred or present with other malignant tumors within 5 years. Patients with the following two conditions can be enrolled: other malignancies treated with a single operation, achieving continuous 5-year disease-free survival (DFS); Cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (cancer in situ) and T1 (tumor infiltrating basal membrane)];
5. Subjects had participated in clinical trials of other antineoplastic drugs within 4 weeks before the group;
6. Has uncontrolled or significant cardiovascular disease.
7. Allergy to any investigational drug or any ingredient or excipient in the drug;
8. Female subjects who are pregnant, lactating or plan to become pregnant during the study.
9. Has any other condition that per protocol or in the opinion of the investigator is inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1039 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (tpCR) rate | At surgery
  The pathological complete response rate described as the absence of invasive tumor cells in the breast and ipsilateral axillary lymph nodes upon microscopic examination following

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Before surgery
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Breast pathological complete response (bPCR) rate | At surgery
  It is defined as no invasive tumor cells in the breast examined by microscopy after primary tumor resection (ypT0/is).
Number of participants with adverse events (AEs) | Assessed every 2 cycles of neoadjuvant therapy prior to surgery, up to approximately 30 days after the last neoadjuvant treatment.
  Assessment of the toxicity profile of regimen according to the National Cancer Institute Common Toxicity Criteria version 5.0 (NCI CTCAE v 5.0).
Identification of HER2-Positive Breast Cancer Molecular Characterization and Subtypes. | Up to approximately 2 years from study enrollment
  Tumor tissue samples are analyzed by gene expression analysis and genome sequencing to classify novel subtypes and compare the molecular characteristics with patients' clinical data.

IPD SHARING:
Plan to Share IPD: No